CLINICAL TRIAL: NCT04284813
Title: Treatment Engagement in Families With Substance Use and Psychosis: A Pilot Study
Brief Title: Families With Substance Use and Psychosis: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Julie McCarthy, Ph.D., Assistant Psychologist, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000220; 1K23DA050808-01 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Psychosis; Substance Use; Substance Use Disorders; Family; Tobacco Use; Nicotine Use Disorder; Cigarette Smoking; Cannabis; Marijuana; Alcohol Use Disorder; Alcohol; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Mental Disorder
Keywords: Family; Substance Use Disorder; Psychosis
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders; Tobacco Use; Tobacco Use Disorder; Cigarette Smoking; Marijuana Abuse; Alcoholism; Schizophrenia; Bipolar Disorder; Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemedicine (Experimental): Community Reinforcement and Family Training for first episode psychosis delivered via telemedicine (CRAFT-FT) with 6-8 weekly sessions of 60-minute therapy.
  Interventions: Behavioral: CRAFT-FT

INTERVENTIONS:
Behavioral: CRAFT-FT — CRAFT-FT will be delivered via telemedicine. Topics include building motivation, self-care, communication, understanding patterns of behavior, positive reinforcement, and negative consequences. The intervention will be tailored to families of individuals experiencing psychosis and substance use who are enrolled in first episode psychosis outpatient services. Participants will be asked to completed assessments at pre-treatment, mid-treatment (approximately week 3), post-treatment, and a follow-up assessment approximately 3 month post-treatment.

SUMMARY:
The purpose of this study is to develop and evaluate an intervention that adapts Community Reinforcement and Family Training (CRAFT) for families experiencing first episode psychosis and substance use delivered via telemedicine (video conferencing). The intervention aims to improve treatment engagement and reduce distress, and it will be delivered via telemedicine (CRAFT-FT). To assess feasibility of the intervention, family members will complete the sessions and provide feedback to refine the treatment manual. Data on client relatives with psychosis will be collected for preliminary assessment purposes. Client relatives will not complete the research study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70.
* Having a relative who:

  1. Is a patient with early course psychosis (DSM-5 schizophrenia, schizoaffective disorder, schizophreniform, psychosis not otherwise specified (NOS), delusional disorder, brief psychotic disorder, major depression with psychosis, and bipolar disorder with psychosis) with first onset in the past 6 years, and
  2. Uses tobacco, alcohol, or cannabis in the past 90 days and/or has no apparent immediate interest in abstinence.
* The person(s) who can best describe the client with psychosis.
* At least 4 days per month contact with the client.
* Access to a computer with internet or mobile phone with video conferencing capabilities.
* Ability to provide written informed consent.
* Speak and read English.

Exclusion Criteria:

* DSM-5 moderate or severe substance use disorder in the past year.
* Lifetime psychotic disorder.
* History of domestic violence with the identified patient (IP).
* Psychiatric, cognitive, or medical impairments that would interfere with the ability to follow through with the treatment plan.

Inclusion Criteria for Client Relatives:

* Ages 18-35.
* First episode psychosis (FEP) onset in the past 6 years with a DSM-5 diagnosis of affective (bipolar disorder or major depressive disorder with psychotic features) or non-affective psychosis (schizophrenia spectrum disorder).

  a. Used tobacco, alcohol, or cannabis within the past 90 days and/or has no apparent immediate interest in abstinence.
* Ability to provide written informed consent.
* Speak/read English

Exclusion Criteria:

* N/A

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie McCarthy, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyers RJ, Miller WR, Hill DE, Tonigan JS. Community reinforcement and family training (CRAFT): engaging unmotivated drug users in treatment. J Subst Abuse. 1998;10(3):291-308. doi: 10.1016/s0899-3289(99)00003-6. PMID 10689661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Family member participant data are reported in the Results Section. Clients with psychosis (n=8) were enrolled for preliminary assessment purposes. They did not complete the intervention, and they have no pre-specified primary or secondary outcome data; thus, no data from client with psychosis are reported in the Results Section.
Period: Overall Study
Arm/Group | Telemedicine
Started | 21 (One family member participant was assigned to the intervention but did not start the intervention due to withdrawal by subject.)
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Family members who started the CRAFT-FT Arm/Group are included in the analyses.
Arm/Group | Telemedicine
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.29 (8.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Sessions Completed
Description: Percentage of sessions completed during the intervention
Time Frame: Post-intervention, approximately Week 6-8
Population: All participants who started the intervention were included in analysis. One family member participant did not start the intervention due to withdrawal by subject.
Measure: Number; unit: percentage of intervention sessions
Arm/Group | Telemedicine
Number analyzed (Participants) | 20
percentage of intervention sessions | 100

2. Secondary Outcome: Mean Session Satisfaction Rating
Description: Participants will report weekly satisfaction ratings following each session on the Session Survey. Ratings will range from 1 (poor) to 5 (excellent) for overall experience and convenience.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemedicine
Number analyzed (Participants) | 20
score on a scale | 4.9 (0.3)

3. Secondary Outcome: Percentage of Participant Preference for In-person, Telemedicine, or Both Session Formats
Description: Percentage of participant preference for in-person, telemedicine, or both sessions formats as assessed categorically during the Treatment Satisfaction Interview.
Time Frame: Up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Telemedicine
Number analyzed (Participants) | 20
Participants
  In-person | 1
  Telemedicine | 9
  Both Session Formate (Hybrid) | 10

ADVERSE EVENTS:
Time Frame: Baseline through 3-month follow-up; 5 months.
Arm/Group | Telemedicine
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemedicine (N=21)
Participant safety concern (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemedicine (N=21)
Cardiac evaluation-hospitalization (Cardiac disorders) | 1 (1) — Unexpected, unrelated.
Interview distress (Psychiatric disorders) | 2 (2) — Expected, related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04284813/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT04284813/ICF_001.pdf